CLINICAL TRIAL: NCT03672994
Title: Exhaled Breath Metabolomic Biomarkers in the Acutely Breathless Patient
Acronym: EMBER
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: Medical Research Council (Other Government); Engineering and Physical Sciences Research Council, UK (Other); Loughborough University (Other); University Hospitals, Leicester (Other); Owlstone Ltd (Industry); B & S ANALYTIK GmbH (Unknown); Advion Biosciences Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0569
Record Dates: First submitted 2018-09-04; First posted 2018-09-17 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2018-08

CONDITIONS: Asthma; COPD; Heart Failure; Community-acquired Pneumonia; Healthy; Breathlessness
Keywords: Acute Breathlessness; Breathomics
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Heart Failure; Community-Acquired Pneumonia; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Asthma: Patients with prior confirmed diagnosis of bronchial asthma
- Chronic Obstructive Pulmonary Disease: Patients with prior confirmed COPD
- Pneumonia: Patients with X-ray confirmed community acquired pneumonia
- Heart failure: Patients with confirmed heart failure
- Healthy volunteers: Healthy participants with no otherwise known cardiorespiratory condition

SUMMARY:
An acute study carried out across three acute admissions units within Leicestershire. The study is aimed at discovery and validation of volatile organic compounds (VOCs) in exhaled breath. Participants will be recruited and tested within 24 hours of admission and once recovered, up to 6 months following discharge.

DETAILED DESCRIPTION:
A prospective real world observational study carried out across three acute admissions units. Participants with self-reported acute breathlessness, with a confirmed primary diagnosis of either acute heart failure, community acquired pneumonia and acute exacerbation of asthma or COPD will be recruited within 24 hours of admission. These will be matched to healthy volunteers from a similar environment. Additionally, school age children admitted with severe asthma will be evaluated and breath samples will be collected. All participants will undergo breath sampling on admission and upon recovery, up to six months following discharge. A range of online technologies including: proton-transfer-reaction mass spectrometry (PTR-MS), gas chromatography ion mobility spectrometry (GC-IMS), atmospheric pressure chemical ionisation- mass spectrometry (APCI-MS) and offline technologies including gas chromatography mass spectroscopy (GC-MS) and comprehensive two-dimensional gas chromatography-mass spectrometry (GCxGC-MS) will be utilised for VOC discovery and replication. For offline technologies a standardised CE marked breath sampling device (ReCIVA®) will be used. All recruited participants will be characterised using existing blood biomarkers including C - reactive protein (CRP), brain derived natriuretic peptide (BNP), Troponin-I and blood eosinophil levels and further evaluated using a range of standardised questionnaires, lung function testing including hand held forced oscillation technique (FOT) and fractional exhaled nitric oxide (FeNO), sputum cell counts and echocardiography for heart failure and COPD patients. Additional samples will be collected for bio-banking including urine, serum, plasma and sputum supernatants and plugs.

ELIGIBILITY:
Inclusion Criteria:

(i) Able to give informed consent for participation in the study. (ii) Male or Female, aged 16 years or above (adult cohort) and 5-15 years for paediatric patients attending the acute care paediatric pathway.

(iii) Capable (in the opinion of the EMBER clinical research investigator(s) of providing serial breath samples.

(iv) Diagnosed with acute breathlessness as one of the primary indicator reasons by the clinical acute care team. This is not a requirement for healthy subjects or matched controls.

(v) One of the indicator provisional diagnoses identified in section 7.1 following senior review by the clinical acute care team. This is not a requirement for healthy subjects or matched controls (vi) Able (in the Investigators opinion) and willing to comply with all study requirements.

(vii) Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

(viii) Ability to understand English.

Exclusion Criteria:

(i) Female participants who are known to be pregnant, lactating or planning pregnancy during the course of the study.

(ii) Current participation in a clinical trial of an investigative medicinal product or within 3 months or 5.5 half-lives of the IMP whichever is longer.

(iii) Active or clinically suspected pulmonary tuberculosis (iv) In the opinion of the treating physician, breath sampling during the acute admission would be clinically unsafe or inappropriate due to the patient's condition or poor prognosis. Examples include malignancy or autoimmune disease with anticipated survival of under 1 year, and chronic renal replacement therapy.

(v) Unable or unwilling to give informed consent by visit 1b. (vi) Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Prospective participants with self reported acute breathlessness, either requiring admission or a change in baseline treatment, presenting within University Hospitals of Leicester (UHL).
  Patients with confirmed acute airway exacerbation or heart failure decompensation as part of other research studies at the NIHR Leicester BRC may also be included.
  Age- and/or home environment matched adult/spousal/parent and sibling healthy volunteers will be recruited where possible on the admissions unit or in the research units across both sites at a separate visit.
  A stable state control population will also be recruited to compare with the unstable state. This will consist of participants with a confirmed diagnosis matched with the acute care population but not in the exacerbation state.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Discovery of exhaled breath biomarkers | 0-6 months
  To evaluate the sensitivity, specificity, positive and negative predictive value of metabolomic biomarkers in exhaled breath samples to identify acute breathlessness, defined as one or more of (i) patient defined acute breathlessness and/or a (ii) 1 unit increase in Extended Medical Research Council breathlessness score (eMRC)

SECONDARY OUTCOMES:
Patient defined breathlessness | visit 1a (first visit), visit 2 (0-6 months)
  Participants are asked to provide information on their state of breathlessness
COPD Assessment Test (CAT) (Questionnaire) | visit 1a (first visit), visit 2 (0-6 months)
  Evaluation and rehabilitation education guidance on the respiratory and motor functions of patients with chronic obstructive pulmonary disease. The CAT has a scoring range of 0-40, with Since COPD is a progressive disease, a fi xed target score for all patients cannot be set. In Practice, a target for improvement in individual patient CAT scores may be set, based on an holistic assessment of the patient. A change of 2 units suggests a meaningful difference. This test should be used in conjunction with the eMRC and forced expiratory volume in one second (FEV1) to determine COPD health assessment of participants.
NASA task load index | visit 1a (first visit), visit 2 (0-6 months)
  Evaluation breath testing work load using mental, physical, temporal, performance, effort and frustration. Participants are asked to mark a scale based on how demanding the task was for each of the domains above.
Asthma quality of life questionaire (AQLQ) | visit 1a (first visit), visit 2 (0-6 months)
  Evaluation quality of life in asthmatic patients based on their level of activity, symptoms, environment and emotion.
Asthma control questionnaire (ACQ) | visit 1a (first visit), visit 2 (0-6 months)
  Measure of asthma control
extended Medical Research Council (eMRC) Dyspnea Scale | visit 1a (first visit), visit 2 (0-6 months)
  Assessing respiratory breathlessness symptoms (Grade 0-5b, with Grade 0 being breathlessness with strenuous exercise to Grade 5b being breathlessness for daily activities like dressing).
Visual analogue score (VAS) total and individual dyspnoea, cough and wheeze (100mm) scores | visit 1a (first visit), visit 2 (0-6 months)
  The participant is asked to place a mark (X) on the scale at the point that best describes their health currently. Minimum score 0mm (better outcome), maximum score 100mm (worse outcome) for each section of the scale (dyspnoea, cough, wheeze).
NewYork Heart Association Dyspnoea score (NYHA) | visit 1a (first visit), visit 2 (0-6 months)
  Assessing grades of breathlessness specifically designed for heart failure patients
Sputum collection for assessment of purulence, cytology and metagenomics | visit 1a (first visit), visit 2 (0-6 months)
  Participants are asked to provide a spontaneous sputum sample assessing purulence, cytology and metagenomics
Pre and post bronchodilator (BD) spirometry to assess lung function | visit 1a (first visit), visit 2 (0-6 months)
  To assess lung function
fraction exhaled nitric oxide (FeNO) assessing airway inflammation | visit 1a (first visit), visit 2 (0-6 months)
  To assess airway inflammation in asthmatics. Patients are asked to blow into a mouthpiece for few seconds which detects the amount of exhaled nitric oxide.
Hand held oscillometry assessing small airway lung function | visit 1a (first visit), visit 2 (0-6 months)
  To assess small airway lung function
Quadriceps ultrasound measuring quadriceps size as a degree of frailty | visit 1a (first visit)
  To assess degree of frailty and muscle breakdown during hospital admission. Participants have their quadriceps muscle size measured using an ultrasound machine.
Four meter gait | visit 1a (first visit), visit 2 (0-6 months)
  physical performance - measure of frailty
Exacerbation history | visit 1a (first visit), visit 2 (0-6 months)
  participants are asked to provide information on recent exacerbations of airway disease
DECAF score assessing in hospital mortality in COPD patients | visit 1a (first visit)
  DECAF score has a minimum score of 1 (better outcome) and a maximum score of 6(worse outcome) used for assessment of severity of COPD exacerbation measures eMRC score, Eosinopenia, consolidation, acidemia and atrial fibrillation
CURB65 score assessing mortality in Pneumonia patients | visit 1a (first visit)
  CURB65 is used in assessment of 30 day mortality of Pneumonia based on confusion, urea, respiratory rate, blood pressure and age.Scores range from 1 (better outcome) to 5 (worse outcome)
BTS asthma severity score | visit 1a (first visit)
  BTS asthma severity score is used in assessment of asthma severity based on peak flow, respiratory rate, oxygen levels, altered level of consciousness, arrythmia, hypotension, cyanosis, silent chest and respiratory effort. Patients are then classified into mild (better outcome), moderate, severe and life threatening (worse outcome).
Meta analysis global group in chronic heart failure (MAGGIC - risk calculator) | visit 1a (first visit)
  Assessment of heart failure severity based on age, gender, diabetes, COPD, heart failure diagnosed in the last 18 months, current smoker, NYHA class, b blockers, ACEI or ARB, BMI, systolic BP, creatinine and ejection fraction
Sputum differential Cell Count | visit 1a (first visit), visit 2 (0-6 months)
  Differential Cell Count to assess inflammation at exacerbation events.
Breath volatile organic compound (VOC) profiling | visit 1a (first visit), visit 2 (0-6 months)
  Participants are asked to provide a breath sample to measure VOC using Compact Mass Spectrometer (CMS), Gas chromatography ion mobility spectrometer (GC-IMS), gas chromatography mass spectrometer (GC-MS), Proton transfer reaction time of flight mass spectrometer (PTR-Tof-MS), gas chromatography gas chromatography mass spectrometer (GCxGC-MS).
Serum/Plasma Inflammatory Biomarkers | visit 1a (first visit), visit 2 (0-6 months)
  To assess systemic inflammation. Plasma/ serum biomarkers are exploratory and we do not have a specific list of biomarkers yet.
Full blood count (FBC) | visit 1a (first visit), visit 2 (0-6 months)
  Blood Biochemistry
C-reactive protein (CRP) | visit 1a (first visit), visit 2 (0-6 months)
  Blood Biochemistry
Troponin-I | visit 1a (first visit), visit 2 (0-6 months)
  Blood Biochemistry
B-type naturitic peptide (BNP) | visit 1a (first visit), visit 2 (0-6 months)
  Blood biochemistry
RNA (PAXgene) | visit 1a (first visit), visit 2 (0-6 months)
  Blood Biochemistry
DNA (PAXgene) | visit 1a (first visit), visit 2 (0-6 months)
  Blood Biochemistry
Age | visit 1a (first visit), visit 2 (0-6 months)
  Demographics
Smoking status, calculated using pack years (no. of cigarettes smoked per day X no. of years smoked divided by 20 | visit 1a (first visit), visit 2 (0-6 months)
  Demographics
BMI in kg/m^2 | visit 1a (first visit), visit 2 (0-6 months)
  Demographics
Gender | visit 1a (first visit), visit 2 (0-6 months)
  Demographics
Heart rate | visit 1a (first visit), visit 2 (0-6 months)
  Vital signs
Blood pressure | visit 1a (first visit), visit 2 (0-6 months)
  Vital signs
Oxygen saturations | visit 1a (first visit), visit 2 (0-6 months)
  Vital signs
Temperature | visit 1a (first visit), visit 2 (0-6 months)
  Vital signs
Medical history | visit 1a (first visit), visit 2 (0-6 months)
  medical history
Current medications | visit 1a (first visit), visit 2 (0-6 months)
  Medical history
Physical examination | visit 1a (first visit), visit 2 (0-6 months)
  Physical examination
12 lead Electrocardiogram (ECG) | visit 1a (first visit), visit 2 (0-6 months)
  cardiac function
Echocardiogram (ECHO) | visit 1a (first visit), visit 2 (0-6 months)
  cardiac function
Chest Xray | visit 1a
  Respiratory function
Height | visit 1a (first visit), visit 2 (0-6 months)
  Demographics
Weight | visit 1a (first visit), visit 2 (0-6 months)
  Demographics
Ethnicity | visit 1a (first visit), visit 2 (0-6 months)
  Demographics
Review of adverse events and serious adverse events | visit 1a (first visit), visit 2 (0-6 months)
  Review of untoward medical occurrences

CONTACTS AND LOCATIONS:
Overall Officials: Salman Siddiqui, Professor, Principal Investigator — University of Leicester
Locations (1):
- NIHR Leicester Biomedical Research Centre - Respiratory, Glenfield Hospital, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ibrahim W, Wilde M, Cordell R, Salman D, Ruszkiewicz D, Bryant L, Richardson M, Free RC, Zhao B, Yousuf A, White C, Russell R, Jones S, Patel B, Awal A, Phillips R, Fowkes G, McNally T, Foxon C, Bhatt H, Peltrini R, Singapuri A, Hargadon B, Suzuki T, Ng LL, Gaillard E, Beardsmore C, Ryanna K, Pandya H, Coates T, Monks PS, Greening N, Brightling CE, Thomas P, Siddiqui S. Assessment of breath volatile organic compounds in acute cardiorespiratory breathlessness: a protocol describing a prospective real-world observational study. BMJ Open. 2019 Mar 8;9(3):e025486. doi: 10.1136/bmjopen-2018-025486. PMID 30852546

DOCUMENTS (2):
  • Study Protocol (2018-04-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT03672994/Prot_000.pdf
  • Informed Consent Form (2018-04-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT03672994/ICF_001.pdf